CLINICAL TRIAL: NCT05307003
Title: Trazodone vs. Quetiapine for the Treatment of ICU Delirium: A Prospective Observational Pilot Study
Brief Title: Trazodone vs. Quetiapine for the Treatment of ICU Delirium
Acronym: TQDelirium
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Catherine Kuza, MD, Assistant Professor of Anesthesiology, University of Southern California
Other Study IDs: HS-22-00540
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Delirium; Delirium of Mixed Origin; Delirium, Sepsis Associated; Delirium in Old Age; Delirium Confusional State; Psych; Morality; Treatment Side Effects
Keywords: critical care; ICU delirium; trazodone; quetiapine; outcomes
MeSH Terms: conditions — Delirium; Sepsis-Associated Encephalopathy; Confusion | interventions — Trazodone; Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Quetiapine: Patients diagnosed with delirium who received quetiapine for treatment.
  * Start study medication at 25 mg daily PO ; may increase to BID (twice a day) or TID (three times a day) if RASS>=2 or rescue medication must be given; thereafter, if med is TID, dose can be increased by increment of 50 mg q12 hr if RASS>=2 and/or >1 dose of rescue medication is given within 24 hours [max dose 200 mg/day]
  * dose can be reduced/discontinued per discretion of ICU attending if delirium improving, patient experiences AE (adverse effects) likely related to study drug, after 14 days of treatment, or patient is discharged from ICU
  * dose should be held if RASS is -3 to -5/comatose/unresponsive or sudden acute change in mental status
  Interventions: Drug: Quetiapine
- Trazodone: Patients diagnosed with delirium who received trazodone for treatment.
  * Start study medication at 25 mg daily PO ; may increase to BID or TID if RASS>=2 or rescue medication must be given; thereafter, if med is TID, dose can be increased by increment of 50 mg q12 hr if RASS>=2 and/or >1 dose of rescue medication is given within 24 hours [max dose 200 mg/day]
  * dose can be reduced/discontinued per discretion of ICU attending if delirium improving, patient experiences AE likely related to study drug, after 14 days of treatment, or patient is discharged from ICU
  * dose should be held if RASS is -3 to -5/comatose/unresponsive or sudden acute change in mental status
  Interventions: Drug: Trazodone

INTERVENTIONS:
Drug: Trazodone — Medication used to treat ICU delirium
  Other Names: Desyrel
  Groups: Trazodone
Drug: Quetiapine — Medication used to treat ICU delirium
  Other Names: Seroquel
  Groups: Quetiapine

SUMMARY:
This is a single-center, prospective observational pilot study. The objective of this study is to evaluate the effectiveness of trazodone as compared to quetiapine, in the management of ICU delirium in adult (>=18 years old) surgical and medical ICU patients. The investigators will compare outcomes such as delirium duration, delirium-free days, coma-free days, in-hospital mortality, 28-day mortality, hospital length of stay (LOS), ICU LOS, mechanical ventilator days, complications, adverse effects, rescue medication use, delirium symptom severity, sleep duration, and sleep quality among participants receiving trazodone or quetiapine. The investigators hypothesize participants receiving trazodone will be associated with a shorter duration of delirium, decreased delirium severity, and improved sleep quality compared to participants receiving quetiapine.

DETAILED DESCRIPTION:
This is a single-center, double-blind randomized, placebo-controlled pilot trial comparing trazodone, quetiapine, and placebo for the treatment of ICU delirium in adult patients admitted to the medical and surgical ICU at Keck Hospital of the University of Southern California.

The purpose of this study is to determine the effectiveness of trazodone and quetiapine for the treatment of ICU delirium, and their effects on patient outcomes. Since the incidence of ICU delirium is high and has profound negative ramifications on survival, long-term outcomes, cognitive function, in addition to placing a heavy burden on the healthcare system resources and costs, effective delirium treatment strategies are desperately needed. Trazodone is a medication that has promise in delirium treatment, but there is currently insufficient literature to recommend its routine use. The investigators' main objective is to determine if trazodone is an effective and safe treatment option for the management of ICU delirium, and if it results in shorter delirium duration and improved outcomes compared to participants receiving quetiapine.

Subject screening:

All patients will be screened for study eligibility daily on rounds throughout the study period. Patients eligible for the study will be enrolled in the study after receiving a patient information sheet. As this is part of standard of care and the medications would be administered regardless of study participation, written informed consent will be waived.

ICU nurses will assess all patients for delirium at least every 12 hours, using the CAM-ICU tool , in accordance with the standard of care in the surgical ICU (that is, this assessment would be performed regardless of the study).

Patients with a diagnosis of delirium (CAM-ICU positive) that requires pharmacological intervention as determined by the attending intensivist, and meet all inclusion criteria and have no exclusion criteria, will receive either trazodone or quetiapine.

Stratification Scheme: Patients who are enrolled in the study, meet inclusion criteria, and have no exclusion criteria, and require a medication intervention for the treatment of ICU delirium, as determined by the attending ICU physician, will be randomized to one of two study arms: 1. Trazodone; or 2. Quetiapine. As an observational study, patients will not be randomized to the intervention. The attending ICU physician will determine which medication to administer to the patient based on their clinical opinion or drug preference.

Study Medication Administration:

The choice of quetiapine or trazodone to treat delirium will be made by the attending intensivist covering the ICU based on their personal preference or the patient's clinical presentation and medical history. The dosage and frequency of either quetiapine or trazodone will also be determined by the prescribing attending intensivist, and will factor in the patient's RASS (Richmond Agitation-Sedation Scale) score and agitation severity. The lowest dosage for both medications is 25 mg, and it may be titrated up and have the frequency adjusted to be administered up to three times a day. The max daily dosage for both medications is 200 mg/day.

The dose of the medications can be reduced/discontinued per discretion of ICU attending if delirium is improving, the patient experiences side effects likely related to study drug, after 14 days of treatment, or if the patient is discharged from ICU.

The dose should be held if RASS is -3 to -5/comatose/unresponsive, or the dose should be decreased if there is increased somnolence.

The decision to stop the medication will be made by the ICU attending, and it should be tapered or discontinued based per the attending intensivists discretion, and should factor in the duration, dosage, and frequency that the patient was receiving the medication.

If the patient is experiencing refractory delirium despite increased doses or frequency of either trazodone or quetiapine, it should be treated per the discretion of the ICU intensivist. Intensivists are encouraged to follow the refractory delirium rescue medication algorithm, described below, however, it is not mandatory. ICU night time coverage is sometimes provided by intensivists who are moonlighting or are not part of the core ICU group, and only cover a night shift once a month, and they may not be familiar with this algorithm. They should administer whatever medications they are comfortable with to immediately control the patient's presenting symptoms. Thus, a standardized delirium rescue medication protocol will not be employed.

Refractory Delirium Rescue Medication Algorithm:

* in event of agitation:

  1. treat pain first (optimize pain management and encourage multimodal therapy [neuraxial/regional techniques, gabapentin (neuroleptics), NSAIDs (if allowed by surgery), lidocaine gtt or patches, acetaminophen, and weak opiates (e.g., tramadol))-avoid ketamine if possible
  2. IV haloperidol 1-10 mg q2hr prn
  3. if still refractory may try olanzapine 5-10 mg PO/SL (sublingual) x1
  4. Still refractory start dexmedetomidine drip 0.2 mcg-1.4 mcg/kg/hr no more than 12 hrs
  5. if patient is intubated and refractory to all of the above, start propofol drip 10mg/hr-80 mg/hr for no more than 12 hrs
  6. May consider adding valproic acid
  7. May consider psychiatric consultation
  8. Add melatonin 5-10 mg qhs to promote sleep hygiene, in addition to steps 1-7
* in event of hallucination:

  1. if patient is not in distress-no additional pharmacological interventions
  2. if patient in distress-may administer IV haloperidol 1-10 mg q2hr prn for short term use (no more than 2 days)

Statistics/Analysis Plan:

-Baseline descriptive statistics: Baseline characteristics of the study population will be presented by treatment group using conventional descriptive statistics, including proportions for categorical variables and means and standard deviations or medians and interquartile ranges for continuous variables, as appropriate based on the data distribution. Comparisons of baseline variables will be performed between treatment groups by two-sample t-test or a non-parametric Wilcoxon rank sum test for continuous variables and chi-square or Fisher's exact tests for categorical variables, as appropriate.

-Analysis of feasibility outcomes: All feasibility outcomes (enrollment rate, delirium incidence among those otherwise eligible, completion of in-hospital and post-discharge outcome assessments) will be summarized as frequencies, with proportions and 95% CIs.

-Analysis of primary efficacy endpoints: The primary outcome is the duration of ICU delirium measured in days. Differences in the duration of delirium between treatment groups will be analyzed by Poisson regression or negative binomial regression if there is evidence of over-dispersion. Patients with delirium episodes lasting less than one day will be classified as 0.5 days. All models will include the medication group (trazodone or quetiapine). Adjusting covariates will include age and initial delirium severity as independent variables. In this observational study, the study medications are not randomized but are assigned by decision of each patient's treating physician. Causal interpretations of the effects of medications on outcomes are therefore weakened to the extent that other patient factors related to outcomes influence the physician's decision to prescribe a particular medication for delirium. We will address this issue by developing propensity scores using a logistic regression model (for administration of trazodone vs quetiapine as the binary dependent variable). Patient factors, including age, delirium severity, sex, and other demographic and clinical factors assessed at baseline prior to administration of study medication will be used as independent variables in the logistic regression model; model coefficients will then be used to quantify a propensity score for each patient. The effect estimate for study treatment will be adjusted using inverse probability weighting, using the propensity score as the weighting variable. Model coefficients will be exponentiated to give the estimated rate ratio for the treatment comparison (trazodone vs quetiapine), with 95% confidence intervals. The referent group for treatment group comparisons will be the quetiapine group (i.e., comparing trazodone to quetiapine).

-Analysis of secondary efficacy endpoints: Secondary outcomes will be evaluated in regression models using inverse probability weighting based on propensity scores as detailed above. Binary secondary endpoints include the proportion of patients with in-hospital mortality, 28-day mortality, 1-month post-discharge mortality, who experience complications, and who use rescue medications. The proportion in each treatment group will be summarized by frequencies (percents) and compared univariately by Fisher's exact test and in a multivariable model by logistic regression. In the logistic regression models, the binary dependent variable will be the particular study outcome (e.g., in-hospital mortality). The primary independent variable of interest will be the study treatment and model covariates will include age and initial delirium severity.

Additional secondary endpoints include the length of hospital stay, length of ICU stay, and duration of mechanical ventilation (if applicable). These outcomes will be analyzed with Poisson or negative binomial regression as described in Section 13.2.3.

Study outcomes that are measured daily (delirium severity measured by CAM-S, nightly sleep duration (hours), number of times awoken at night, and sleep quality (Richards Campbell Sleep Questionnaire) will be compared among treatment groups using generalized linear mixed effects models (GLMMs). Normally distributed continuous outcomes will use a normal random outcome with an identify link function; count outcomes (e.g., number of times awoken) will use a Poisson random variable with a log link function. For each model, the primary independent variables will be study treatment group, age, and initial delirium severity. Assessment time (day of assessment, from day 0 to 14) will be treated as indicator variables. The main effect of treatment will estimate and test differences in the mean of the outcome in each study medication group over the 14-day follow-up period. An interaction term of treatment-by-day will be used to estimate treatment group means (with standard errors (SEs) and confidence intervals) by intervention day.

-Analysis of safety measures: Numbers and percentages of adverse events and serious adverse events will be tabulated and summarized descriptively (as frequency and percent, with 95% CI) by treatment group. Major safety measures of interest will be the occurrence of prolonged QTc intervals, extrapyramidal symptoms and muscle rigidity. The two treatment groups will be compared on the proportions exhibiting these adverse effects by Fisher's exact tests.

-Populations for analysis: The full analysis dataset will be comprised of all study participants who have met study inclusion criteria, and been treated with either trazodone or quetiapine. Analysis will be based on the original intervention, regardless of actual intervention received.

ELIGIBILITY:
Inclusion Criteria:

* >=18-years-old
* Admitted to the surgical ICU for >24 hours
* Diagnosis of ICU delirium defined by positive CAM-ICU score AND exhibiting symptomatic delirium (i.e., combative, pulling at lines, a danger to self or others, inability to sleep, hallucinations, etc.), thus, requiring the need for pharmacologic intervention as determined by the attending intensivist
* Receiving either quetiapine or trazodone for the treatment of delirium

Exclusion Criteria:

* Presence of an acute neurologic condition (i.e., acute cerebrovascular accident, intracranial tumor, traumatic brain injury, etc.) on ICU admission. History of stroke or other neurological condition(s) without cognitive impairment is not an exclusion criterion.
* Pregnancy/lactation
* History of ventricular arrhythmia including torsade de pointes or second- and third-degree heart block
* Allergy/hypersensitivity reaction to trazodone and/or quetiapine
* Diagnosis of dementia
* History of neuroleptic malignant syndrome and/or serotonin syndrome
* Diagnosis of Parkinson's disease or parkinsonism (also referred to as hypokinetic rigidity syndrome)
* Schizophrenia or other psychotic disorder
* Patients in whom CAM-ICU cannot be performed to screen for delirium (i.e., acute encephalopathy, mental retardation, vegetative state, deaf, blind, etc.) [reversible coma (that is, not caused by traumatic brain injury, cerebrovascular accident, or intracranial tumor), defined as RASS -4 or -5 at any point through one ICU day, is NOT an exclusion criterion.]
* Inability to speak or understand English
* Expected to die or transfer out of the ICU within 24 hours
* Acute alcohol or substance abuse withdrawal symptoms/syndrome (i.e., delirium tremens) requiring treatment/intervention (e.g, implementation of the Clinical Institute Withdrawal Assessment for Alcohol (CIWA) protocol, benzodiazepines, alpha-2 agonist, etc.)
* Prolonged QTc syndrome AND/OR prolonged QT-interval (QTc>450 ms for men, and >460 ms for women on ECG performed within 1 month of ICU admission or day of study enrollment)
* Active psychosis [defined as distortion or loss of contact with reality, delusions and/or
* hallucinations (without insight), and/or thought disorder-must be diagnosed by a psychiatrist]
* Patients taking medications with known interactions with either trazodone and/or quetiapine per Pharmacy (e.g., MAOIs (monoamine oxidase inhibitors), SSRIs (selective serotonin reuptake inhibitors; etc.)
* Acute encephalopathy (i.e., hepatic, uremic, etc.)
* Seizure disorder
* Myocardial infarction (MI) within the past 30 days
* Tardive dyskinesia
* Symptomatic hyponatremia
* Terminal state
* Diagnosis of liver disease
* Patients who are strict NPO (nil per os), are a high aspiration risk (defined as frequent nausea/vomiting, ileus, gastric dysmotility disorder, uncontrolled gastroesophageal reflux disease, weakness/deconditioning, diabetes with gastroparesis, not tolerating full tube feeds if being enterally fed (high residual gastric volume >500 cc), elderly patients with waxing/waning mental status), have dysphagia, and/or have difficulty swallowing capsules or solutions as determined by speech therapist
* Currently enrolled and participating in another interventional study
* Patients who have received both trazodone and quetiapine in the management of their delirium
* Patients who have had a history of serotonin syndrome
* Patients who were enrolled in the study once, are not eligible for re-enrollment if they are readmitted to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the medical or surgical ICU for >24 hours with delirium requiring treatment with either trazodone or quetiapine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
delirium duration using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) tool | 14 days
  days
delirium-free days | 14 days
  days
coma-free days | 14 days
  days

SECONDARY OUTCOMES:
in-hospital mortality | 365 days
  yes or no
ICU length of stay | 14 days
  days
total hospital length of stay | 14 days
  days
mechanical ventilator days | 14 days
  days
28-day mortality | 28 days
  yes or no
complications | 14 days
  yes or no
adverse effects of study drugs | 14 days
  yes or no
use of rescue medications | 14 days
  yes or no
delirium severity | 14 days
  Confusion Assessment Method-Severity (CAM-S) long form [0= minimum; 19=maximum; increase in score means worse outcome]
sleep quality | 14 days
  using Richards Campbell Sleep Questionnaire
post-discharge depression | 1-month post-hospital discharge
  measured using Hospital Anxiety and Depression Scale [ 0=minimum;21=maximum; the higher the score the higher the chance of depression and worse outcome]
post-discharge anxiety | 1-month post-hospital discharge
  measured using Hospital Anxiety and Depression Scale [ 0=minimum;21=maximum; the higher the score the higher the chance of anxiety and worse outcome]

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Kuza, MD, FASA, Principal Investigator — Keck School of Medicine of the University of Southern California
Locations (1):
- Keck Hospital of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson P, Khan A. Delirium in critically ill patients. Crit Care Clin. 2015 Jul;31(3):589-603. doi: 10.1016/j.ccc.2015.03.011. Epub 2015 May 4. PMID 26118922
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Salluh JI, Latronico N. Making advances in delirium research: coupling delirium outcomes research and data sharing. Intensive Care Med. 2015 Jul;41(7):1327-9. doi: 10.1007/s00134-015-3864-4. Epub 2015 Jun 3. No abstract available. PMID 26077062
- [Background] Zhang H, Lu Y, Liu M, Zou Z, Wang L, Xu FY, Shi XY. Strategies for prevention of postoperative delirium: a systematic review and meta-analysis of randomized trials. Crit Care. 2013 Mar 18;17(2):R47. doi: 10.1186/cc12566. PMID 23506796
- [Background] Ringdal GI, Ringdal K, Juliebo V, Wyller TB, Hjermstad MJ, Loge JH. Using the Mini-Mental State Examination to screen for delirium in elderly patients with hip fracture. Dement Geriatr Cogn Disord. 2011;32(6):394-400. doi: 10.1159/000335743. Epub 2012 Feb 1. PMID 22301509
- [Background] Roberts DJ, Goralski KB, Renton KW, Julien LC, Webber AM, Sleno L, Volmer DA, Hall RI. Effect of acute inflammatory brain injury on accumulation of morphine and morphine 3- and 6-glucuronide in the human brain. Crit Care Med. 2009 Oct;37(10):2767-74. doi: 10.1097/CCM.0b013e3181b755d5. PMID 19865006
- [Background] Collinsworth AW, Priest EL, Campbell CR, Vasilevskis EE, Masica AL. A Review of Multifaceted Care Approaches for the Prevention and Mitigation of Delirium in Intensive Care Units. J Intensive Care Med. 2016 Feb;31(2):127-41. doi: 10.1177/0885066614553925. Epub 2014 Oct 27. PMID 25348864
- [Background] van den Boogaard M, Schoonhoven L, Evers AW, van der Hoeven JG, van Achterberg T, Pickkers P. Delirium in critically ill patients: impact on long-term health-related quality of life and cognitive functioning. Crit Care Med. 2012 Jan;40(1):112-8. doi: 10.1097/CCM.0b013e31822e9fc9. PMID 21926597
- [Background] Davydow DS. Symptoms of depression and anxiety after delirium. Psychosomatics. 2009 Jul-Aug;50(4):309-16. doi: 10.1176/appi.psy.50.4.309. PMID 19687169
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Kamdar BB, King LM, Collop NA, Sakamuri S, Colantuoni E, Neufeld KJ, Bienvenu OJ, Rowden AM, Touradji P, Brower RG, Needham DM. The effect of a quality improvement intervention on perceived sleep quality and cognition in a medical ICU. Crit Care Med. 2013 Mar;41(3):800-9. doi: 10.1097/CCM.0b013e3182746442. PMID 23314584
- [Background] Reznik ME, Slooter AJC. Delirium Management in the ICU. Curr Treat Options Neurol. 2019 Nov 14;21(11):59. doi: 10.1007/s11940-019-0599-5. PMID 31724092
- [Background] Marra A, Ely EW, Pandharipande PP, Patel MB. The ABCDEF Bundle in Critical Care. Crit Care Clin. 2017 Apr;33(2):225-243. doi: 10.1016/j.ccc.2016.12.005. PMID 28284292
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Michaud CJ, Bullard HM, Harris SA, Thomas WL. Impact of Quetiapine Treatment on Duration of Hypoactive Delirium in Critically Ill Adults: A Retrospective Analysis. Pharmacotherapy. 2015 Aug;35(8):731-9. doi: 10.1002/phar.1619. Epub 2015 Aug 4. PMID 26238778
- [Background] Mangan KC, McKinzie BP, Deloney LP, Leon SM, Eriksson EA. Evaluating the risk profile of quetiapine in treating delirium in the intensive care adult population: A retrospective review. J Crit Care. 2018 Oct;47:169-172. doi: 10.1016/j.jcrc.2018.07.005. Epub 2018 Jul 5. PMID 30005303
- [Background] Devlin JW, Roberts RJ, Fong JJ, Skrobik Y, Riker RR, Hill NS, Robbins T, Garpestad E. Efficacy and safety of quetiapine in critically ill patients with delirium: a prospective, multicenter, randomized, double-blind, placebo-controlled pilot study. Crit Care Med. 2010 Feb;38(2):419-27. doi: 10.1097/CCM.0b013e3181b9e302. PMID 19915454
- [Background] Devlin JW, Skrobik Y, Riker RR, Hinderleider E, Roberts RJ, Fong JJ, Ruthazer R, Hill NS, Garpestad E. Impact of quetiapine on resolution of individual delirium symptoms in critically ill patients with delirium: a post-hoc analysis of a double-blind, randomized, placebo-controlled study. Crit Care. 2011;15(5):R215. doi: 10.1186/cc10450. Epub 2011 Sep 17. PMID 21923923
- [Background] Knauert MP, Haspel JA, Pisani MA. Sleep Loss and Circadian Rhythm Disruption in the Intensive Care Unit. Clin Chest Med. 2015 Sep;36(3):419-29. doi: 10.1016/j.ccm.2015.05.008. Epub 2015 Jun 29. PMID 26304279
- [Background] Madrid-Navarro CJ, Sanchez-Galvez R, Martinez-Nicolas A, Marina R, Garcia JA, Madrid JA, Rol MA. Disruption of Circadian Rhythms and Delirium, Sleep Impairment and Sepsis in Critically ill Patients. Potential Therapeutic Implications for Increased Light-Dark Contrast and Melatonin Therapy in an ICU Environment. Curr Pharm Des. 2015;21(24):3453-68. doi: 10.2174/1381612821666150706105602. PMID 26144941
- [Background] Pulak LM, Jensen L. Sleep in the Intensive Care Unit: A Review. J Intensive Care Med. 2016 Jan;31(1):14-23. doi: 10.1177/0885066614538749. Epub 2014 Jun 10. PMID 24916753
- [Background] Okamoto Y, Matsuoka Y, Sasaki T, Jitsuiki H, Horiguchi J, Yamawaki S. Trazodone in the treatment of delirium. J Clin Psychopharmacol. 1999 Jun;19(3):280-2. doi: 10.1097/00004714-199906000-00018. No abstract available. PMID 10350040
- [Background] Popeo DM. Delirium in older adults. Mt Sinai J Med. 2011 Jul-Aug;78(4):571-82. doi: 10.1002/msj.20267. PMID 21748745
- [Background] Wada K, Morita Y, Iwamoto T, Mifune Y, Nojima S. First- and second-line pharmacological treatment for delirium in general hospital setting-Retrospective analysis. Asian J Psychiatr. 2018 Feb;32:50-53. doi: 10.1016/j.ajp.2017.11.028. Epub 2017 Dec 5. PMID 29216606
- [Background] Maeda I, Inoue S, Uemura K, Tanimukai H, Hatano Y, Yokomichi N, Amano K, Tagami K, Yoshiuchi K, Ogawa A, Iwase S; Phase-R Delirium Study Group. Low-Dose Trazodone for Delirium in Patients with Cancer Who Received Specialist Palliative Care: A Multicenter Prospective Study. J Palliat Med. 2021 Jun;24(6):914-918. doi: 10.1089/jpm.2020.0610. Epub 2021 Feb 11. PMID 33577386
- [Background] Berman BD. Neuroleptic malignant syndrome: a review for neurohospitalists. Neurohospitalist. 2011 Jan;1(1):41-7. doi: 10.1177/1941875210386491. PMID 23983836
- [Background] Scotton WJ, Hill LJ, Williams AC, Barnes NM. Serotonin Syndrome: Pathophysiology, Clinical Features, Management, and Potential Future Directions. Int J Tryptophan Res. 2019 Sep 9;12:1178646919873925. doi: 10.1177/1178646919873925. eCollection 2019. PMID 31523132
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Hodgson C, Needham D, Haines K, Bailey M, Ward A, Harrold M, Young P, Zanni J, Buhr H, Higgins A, Presneill J, Berney S. Feasibility and inter-rater reliability of the ICU Mobility Scale. Heart Lung. 2014 Jan-Feb;43(1):19-24. doi: 10.1016/j.hrtlng.2013.11.003. Epub 2013 Nov 19. PMID 24373338
- [Background] Jones C, Griffiths RD, Humphris G, Skirrow PM. Memory, delusions, and the development of acute posttraumatic stress disorder-related symptoms after intensive care. Crit Care Med. 2001 Mar;29(3):573-80. doi: 10.1097/00003246-200103000-00019. PMID 11373423
- [Background] Breitbart W, Gibson C, Tremblay A. The delirium experience: delirium recall and delirium-related distress in hospitalized patients with cancer, their spouses/caregivers, and their nurses. Psychosomatics. 2002 May-Jun;43(3):183-94. doi: 10.1176/appi.psy.43.3.183. PMID 12075033
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ishii T et al. Retrospective Study of Trazodone Monotherapy Compared with Ramelteon and Trazodone Combination Therapy for the Management of Delirium. J Psychiatry. 2018; 21(3):1-5
- [Background] Ospina JP et al. Epidemiology, Mechanisms, Diagnosis, and Treatment of Delirium: A Narrative Review. Clinical Medicine and Therapuetics. 2018;1(1):3-9.